CLINICAL TRIAL: NCT00212186
Title: Selenium Supplementation of Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, RBurk, M.D., Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DK54819; R01DK058763 (NIH); 1R03DK054819 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Healthy; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

INTERVENTIONS:
Drug: Selenium Supplements (essential nutrient)

SUMMARY:
The purpose of this study is to determine whether patients with liver disease can improve their nutritional selenium status by taking supplemental selenium.

DETAILED DESCRIPTION:
Selenium is an essential nutrient. Selenium carries out its biological functions through selenoproteins. The most abundant selenoprotein in the plasma is selenoprotein P, which is largely synthesized in the liver. Patients with liver disease often have less than half the selenoprotein P levels of normal individuals. This suggests that people with liver disease are not meeting their selenium requirements and may benefit from additional selenium.

We proposed to compare the effects of two different forms of supplemental selenium on plasma selenium levels among patients with severe liver cirrhosis and healthy individuals (controls). Patients and controls were randomly assigned to one of 3 treatment groups: 200 µg selenium per day as selenate, 200 µg selenium per day as selenomethionine, or a placebo. The intervention lasted 8 weeks. Blood was measured initially and after 2 and 4 weeks of supplementation. Selenium, selenoprotein P and glutathione peroxidase were measured in the plasma. We compared changes in selenium and selenoprotein levels between liver cirrhosis patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults
* Adults with Child-Pugh Class C liver cirrhosis

Exclusion Criteria:

* Diagnosis of renal failure
* Urgent need of liver transplant
* Selenium supplements of >25 µg per day during the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1998-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Plasma Selenium Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Burk, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States